CLINICAL TRIAL: NCT04288505
Title: Evaluation of a Virtual Reality Tool for Identifying the Cognitive Functions of the Right Hemisphere in Patients With Brain Damage -TANGO
Acronym: TANGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A00074-35
Record Dates: First submitted 2020-02-14; First posted 2020-02-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Virtual Reality; Brain Damage
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental)
  Interventions: Diagnostic Test: VIRTUAL REALITY application

INTERVENTIONS:
Diagnostic Test: VIRTUAL REALITY application — application on virtual reality headset

SUMMARY:
Evaluate the diagnostic performance of a virtual reality application to detect the presence of cognitive impairment of the non-dominant hemisphere in patients with brain damage

ELIGIBILITY:
Inclusion Criteria:

* Indication for brain lesion located in the right hemisphere surgery
* Major patient
* Karnofsky ≥ 70

Exclusion Criteria:

* Person with aphasia
* Person with visual problems
* Person with a contraindication to MRI
* Person unable to carry out the tests planned in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Performance of the virtual reality application compared to classic cognitive tests batery for the detection of cognitive deficit | from surgery to 3 months after surgery

SECONDARY OUTCOMES:
Performance of the virtual reality application compared with conventional cognitive tests used to detect visual-spatial attention disorders | from surgery to 3 months after surgery
Performance of the virtual reality application compared with conventional cognitive tests used to detect facial emotion recognition disorders | from surgery to 3 months after surgery
Performance of the virtual reality application compared with conventional cognitive tests, used to detect spatial attention disorders or the presence of facial emotion recognition disorders depending respectively on the location or type of facial emotion | from surgery to 3 months after surgery
Study the reproducibility of the virtual reality application for detecting the presence of cognitive function disorders | from surgery to 3 months after surgery
Study the correlation between visuo-spatial and facial emotion recognition deficits and possible tractographic changes | from surgery to 3 months after surgery
Study the association between the presence of cognitive function deficits and the presence of behavioral disorders or health-related quality of life | from surgery to 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No